CLINICAL TRIAL: NCT01278381
Title: A PROGNOSTIC SCORE TO PREDICT MAJOR COMPLICATIONS AFTER PANCREATICODUODENECTOMY.
Brief Title: Prognostic Score To Predict Major Complications After Pancreaticoduodenectomy
Status: Completed | Type: Observational
Sponsor: Università Vita-Salute San Raffaele (Other)
Responsible Party: Marco Braga, MD, Università Vita-Salute San Raffaele
Other Study IDs: PANCREATICODUODENECTOMY_SCORE
Record Dates: First submitted 2011-01-14; First posted 2011-01-17 (Estimated); Last update posted 2011-01-17 (Estimated); Status verified 2010-11

CONDITIONS: Pancreatic Neoplasm
Keywords: pancreas, pancreaticoduodenectomy, major complications
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Pancreaticoduodenectomy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Pancreaticoduodenectomy (PD): Patients undergoing PD from 2002 to 2010
  Interventions: Procedure: Pancreaticoduodenectomy

INTERVENTIONS:
Procedure: Pancreaticoduodenectomy — Resection of pancreatic lesion

SUMMARY:
Pancreaticoduodenectomy (PD) still carries a high rate of severe postoperative complications. No score is currently available to help identify the patient's surgical risk. The purpose of this study was to develop and validate a prognostic score to predict major postoperative complications after PD.

DETAILED DESCRIPTION:
The investigators prospectively collected in an electronic database preoperative, intraoperative and outcome data of 700 patients undergoing PD in our Institution from 2002 to 2010. The investigators used a multivariate logistic regression analysis to create a new score to predict severe complications defined as Clavien-Dindo classification III, IV and V. The score was developed using a random two-thirds of the population (469 patients), and was then validated and calibrated in the remaining third of the patients (231).

ELIGIBILITY:
Inclusion Criteria:

- Patients undergoing pancreaticoduodenectomy in our Institution

Exclusion Criteria:

* Metastatic disease
* Patient not suitable for surgery

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 700 patients undergoing pancreaticoduodenectomy in our Institution from 2002 to 2010
Sampling Method: Non-Probability Sample
Enrollment: 700 (Actual)
Dates: Start 2002-01; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
Major Complication rate | Postoperative. Until 30 days after discharge
  Clavien-Dindo grade III to V complications considered as major

CONTACTS AND LOCATIONS:
Overall Officials: Marco Braga, MD, Principal Investigator — Università Vita-Salute San Raffaele
Locations (1):
- San Raffaele Hospital, Milan, Italy